CLINICAL TRIAL: NCT07356882
Title: Non-interventional Research Protocol Involving Human Participants
Brief Title: European Project for ctDNA Detection as a Biomarker for Non-invasive Therapy Monitoring in Paediatric Classical Hodgkin Lymphoma
Acronym: EURHOLY
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre de Lutte contre le Cancer Henri Becquerel, Rouen, France (Unknown); University Medical Center of Giessen, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP241626; IDRCB 2025-A01092-47 (Other: ANSM)
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: Classical Hodgkin lymphoma; Pediatric oncology; Circulating tumor DNA (ctDNA); Liquid biopsy; Risk stratification; Minimal residual disease (MRD); Biomarker; Next-Generation Sequencing (NGS); Treatment response evaluation; Relapse prediction; PET/CT correlation
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Cohort: ctDNA analysis at 4 timepoints during standard treatment

SUMMARY:
Classical Hodgkin lymphoma (cHL) accounts for 15% of all cases of cancer in children and adolescents and represents the first cause of cancer during adolescence. Combined multi-modal chemotherapy and modern radiation techniques have transformed cHL in a highly curable cancer. However, up to 10-15% of patients still experience recurrent or primary refractory disease. Thus, there is an unmet need for unravelling the underlying mechanisms of treatment failure and refractoriness in paediatric cHL. Further refinements of treatment strategy are still needed to improve treatment results both in relapse and refractory (R/R) patients and to reduce long-term morbidity and mortality treatment related. Therefore, two main objectives arise: to improve early detection of patients with a high relapse risk to potentially intensify the first line treatment and to better identify low risk patients to further reduce the treatment burden in this good-prognostic population. Initial disease stratification and long-term outcome predictions remain a challenging issue in the field. PET/CT is currently the reference imaging method for initial staging and improves detection of extra nodal disease. None of previous prognostic factors accurately identify patients who will respond adequately and therefore limit the ability to identify patients who should require treatment that is more intensive or new therapeutic approaches like immunotherapy. Taken together, these data emphasize a clear unmet need in the field of cHL. We aim to develop a biomarker tool, which could sharpen the initial risk stratification, improve the assessment of disease evaluation during the treatment and beyond and facilitate the detection of relapse. Over the past decade, as in other malignancies the potential of quantification of circulating tumour DNA (ctDNA) or liquid biopsy, in circulating cell-free DNA (cfDNA) that comprises DNA fragments released from apoptotic or necrotic cells into circulation, has emerged as a promising tool for diagnosis and exploration of the genetic landscape associated with HRS and for response evaluation. Experiences of ctDNA in cHL was first reported in adult cHL. These previous studies paved the way for ctDNA implementation in cHL. First, they contributed to confirm the feasibility to use ctDNA in the detection of tumor-associated mutation. Using paired samples of ctDNA and tumor DNA from HRS cells obtained by microdissection they confirmed the consistent correlation between these two methods. Second, they highlighted the potential role of ctDNA as a surrogate marker for tumor baseline assessment and more importantly for interim evaluation reporting an excellent correlation between the PET/CT result and the presence or the absence of ctDNA after 2 cycles of chemotherapy. Furthermore, Sobesky et al. previously reported that cured patients who were inconsistently judged as interim PET/CT-positive had a more than 2-log drop in ctDNA, whereas relapsing patients who were inconsistently judged as interim PET/CT negative had a less than 2-log drop in ctDNA. These data suggest that ctDNA could be a relevant adjunct to conventional PET/CT approach.

DETAILED DESCRIPTION:
Despite significant advances in the management of classical Hodgkin lymphoma (cHL) in children and adolescents, a proportion of patients still relapse or exhibit primary refractory disease. This highlights a persistent limitation in current prognostic tools, particularly in identifying, at diagnosis or early during treatment, those at high risk of treatment failure. Existing stratification systems rely on clinical features and PET/CT imaging, which, although valuable, do not consistently differentiate between patients requiring intensification and those who could benefit from treatment de-escalation.

To address this unmet need, the use of circulating tumor DNA (ctDNA) as a non-invasive biomarker has emerged as a promising avenue. ctDNA analysis allows real-time molecular assessment of tumor dynamics, including mutation detection and disease burden, without requiring invasive tissue biopsies. In adult cHL, ctDNA has demonstrated feasibility, prognostic relevance, and strong correlation with PET/CT results during treatment. Its early kinetics may even outperform imaging in predicting treatment outcomes, particularly in discordant PET scenarios.

In pediatric cHL, ctDNA remains underexplored. The HOLY study, a French initiative nested within the EuroNet-PHL-C2 framework, was among the first to evaluate ctDNA detection in this population using a targeted panel of 18 recurrently mutated genes. Preliminary findings show a high mutation detection rate (~85%) in baseline plasma samples. Parallel efforts in Germany (PHL-ctDNA study) use a broader panel and an alternative detection method, offering a valuable opportunity for methodological comparison and data integration.

The current study proposes a binational collaborative approach involving France and Germany to:

* Extend and harmonize ctDNA analyses in pediatric cHL;
* Compare sequencing methodologies for sensitivity, specificity, and clinical concordance;
* Integrate ctDNA dynamics with imaging and clinical outcomes to refine prognostic models.

This will culminate in a prospective trial using a unified NGS panel (~80 genes), informed by pooled retrospective analysis. ctDNA will be assessed at strategic timepoints to evaluate its added value in relapse prediction and risk-adapted therapy.

Ultimately, this work seeks to validate ctDNA as a central biomarker for early response assessment, molecular monitoring, and personalized treatment planning in pediatric cHL.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed classical Hodgkin lymphoma (cHL)
* Children and young adults under the age of 25 years old
* Signature of informed consent by the patient and/or holders of parental authority (depending on the age of the patient)
* Affiliation to a social security scheme or being beneficiary of such a scheme

Exclusion Criteria:

* Previous treatment with chemotherapy or radiotherapy for another cancer
* Pretreatment of Hodgkin lymphoma (except one treatment with corticosteroid for 7 to 10 days for large or compressive mediastinal tumors).
* Diagnosis of nodular lymphocyte predominant Hodgkin lymphoma (NLPHL)
* Other concomitant malignancies • Residence outside participating countries in for which long-term follow-up cannot be ensured

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adolescents newly diagnosed with Hodgkin lymphoma treated in participating pediatric oncology centers. Patients will be enrolled at diagnosis and followed prospectively for relapse outcomes
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival (RFS) at 2 and 5 years based on ctDNA status at diagnosis | 2 years and 5 years
  Time from initial diagnosis to first relapse or death from any cause. Patients will be stratified by ctDNA status at diagnosis, including quantitative burden and mutation profiles.

SECONDARY OUTCOMES:
Diagnostic performance of ctDNA after 1 cycle of chemotherapy | At Day 28 (post first OEPA cycle)
  Sensitivity, specificity, PPV and NPV of ctDNA detection compared to PET/CT metrics (deltaSUVmax, Deauville score).
Diagnostic performance of ctDNA after 2 cycles of chemotherapy | At Day 56 (post second OEPA cycle)
  Sensitivity, specificity, PPV and NPV of ctDNA detection compared to PET/CT metrics (deltaSUVmax, Deauville score).
Diagnostic performance of ctDNA at end of treatment | At treatment completion (approximately Month 6)
  Sensitivity, specificity, PPV and NPV of ctDNA detection at end of treatment compared to PET/CT evaluation.
Molecular landscape of ctDNA at relapse | Up to 5 years
  Mutation profiling of ctDNA in patients with relapsed/refractory cHL and analysis of association between mutation patterns and treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu SIMONIN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pediatric Hematology and Oncology Department, Paris, France